CLINICAL TRIAL: NCT00638027
Title: Memantine for Spasticity in MS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Andrew Goodman, MD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8049
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Memantine 10 mg bid
  Interventions: Drug: memantine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — matched tablets bid
  Arms: 2
Drug: memantine — 10 mg bid
  Other Names: Namenda
  Arms: 1

SUMMARY:
Participants (n=20) will be identified at routine care visits performed at the Rochester Multiple Sclerosis Center. Eligible participants will have MS by McDonald Criteria,7 and will have a modified Ashworth spasticity rating8 of two or higher in at least one lower extremity muscle group. Participants will be seen at screening, one, and three months, and will be evaluated using the modified Ashworth scale,8 pendulum test,9 toe tapping test,10 manual muscle testing,11 timed 25 foot walk,12 and Multiple Sclerosis Functional Composite.13 The type and severity of any adverse events will be recorded using standard definitions. Participants will be instructed to call between visits to inform the investigators regarding any adverse events they experience. Follow-up will continue until all adverse events resolve or stabilize.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, double-blind, parallel group trial of memantine in patients with MS and spasticity. Participants will be identified at routine care visits at the Rochester Multiple Sclerosis Center. After obtaining informed consent, patients will undergo screening, which will include a physical/neurologic exam and an assessment of the Expanded Disability Status Scale, spasticity, and functional abilities. Eligible patients will return for a baseline evaluation, will initiate their randomly assigned study medication, and will return after one and three months for re-evaluation. The type and severity of any adverse events will be recorded using standard definitions. Participants will be instructed to call between visits to inform the investigators regarding any adverse events they experience. Follow-up will continue until all adverse events resolve or stabilize.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple sclerosis by McDonald Criteria.
2. Spasticity. A minimum score of two on the Ashworth spasticity scale in at least one lower extremity muscle group and a total score of at least four in the lower extremity muscles tested.
3. Age 18-70.
4. Normal renal function (estimated CrCl > 50 ml/min).
5. Women of childbearing potential (i.e., those not postmenopausal or surgically sterile) may participate provided that they are using adequate birth control methods (including barrier methods, IUD, and oral contraceptives) for the duration of the study.
6. Willing and able to perform all procedures related to the clinical trial and to provide informed consent.

Exclusion Criteria:

1. Evidence of clinically significant thyroid, gastrointestinal, cardiovascular, hepatic, renal, hematologic, respiratory, neoplastic, endocrine (including diabetes mellitus), neurologic (other than MS), or other medical or psychiatric disorder at screening.
2. Women must not be pregnant or lactating. Serum or urine pregnancy tests will be required prior to randomization for women of childbearing potential unless the last menstrual period started less than 28 days prior to randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Goodman, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Mehta LR, McDermott MP, Goodman AD, Schwid SR. A randomized trial of memantine as treatment for spasticity in multiple sclerosis. Mult Scler. 2010 Feb;16(2):248-51. doi: 10.1177/1352458509355462. Epub 2009 Dec 22. PMID 20028712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the trial began in June 2006 and ended in June 2008. The last subject formally completed the trial in September 2008
Groups:
- Memantine: Memantine 10 mg bid
- Placebo: Placebo arm
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 11 | 10
Completed | 11 | 8 (all 10 included in analyses)
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (7.5) | 52.1 (12.2) | 52.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Difference in Ashworth Spasticity Scale Score Between Baseline and 12 Weeks
Description: spasticity scale score: the most common used tool to measure the degree of spasticity of the lower extremities.
  Score: Degree of Muscle Tone 0: no increase in tone
  1. slight increase in tone 1+: slight increase in tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion.
  2. more marked increase in muscle tone through most of the range of movement, but affected part(s) easily moved.
  3. considerable increase in muscle tone, passive movement difficult.
  4. affected part(s) rigid in flexion or extension.
Time Frame: Baseline and 12 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | -1.55 (2.81) | -1.00 (2.67)

2. Secondary Outcome: Difference in the Multiple Sclerosis Spacticy Scale (MSSS-88) Between Baseline and 12 Weeks
Description: Multiple Sclerosis Spacticy Scale (MSSS-88) is a patient reported questionnaire rating scale to quantify the perspectives of the impact of spasticity on people with multiple sclerosis.
  Scoring: Individual items are scored on a 4 point Likert scale: 1 (Not bothered at all), 2 (a little bothered), 3 (moderately bothered), 4 (extremely bothered).This questionnaire asks how bothered you have been by your spasticity in the past two weeks. By spasticity we mean muscle stiffness and spasms.The MSSS-88 is a reliable and valid, patient-based, interval-level measure of the impact of spasticity in multiple sclerosis. Scores were summed, without weighting or standardization, to generate ordinal-level total scores just as any other Likert-type scale. Missing responses to items can be replaced with the mean score of the items completed (person-specific item mean score) provided that 50% or more of the items in a scale have been completed. The range is 8-32 and higher scores mean poorer outcome.
Time Frame: baseline, 12 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | -5.55 (7.89) | -3.33 (7.07)

3. Secondary Outcome: Change in Multiple Sclerosis Functional Composite (MSFC) Score Between Baseline and Week 12
Description: 9-Hole Peg Test (9-HPT) is a quantitative measure of upper extremity function. Timed 25-Foot Walk (T 25 FW) is a quantitative measure of lower extremity function. The patient is instructed to walk 25 feet as quickly as possible, but safely.
  Paced Auditory Serial Addition Test-3 seconds (PASAT-3) is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability.
  The MSFC is based on the concept that scores for these 3 dimensions-arm, leg, and cognitive function are combined to create a single score that can be used to detect change over time in a group of MS patients. This is done by creating Z-scores for each component of the MSFC. Implicit in this approach is the idea that patients who deteriorate or improve on all 3 component measures will have an overall larger change than patients who change on only 1 of the 3 measures. The MSFC score was transformed to z-scores, with higher scores indicating better outcome.
Time Frame: Baseline, Week 12
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 10
Z score | 0.02 (0.26) | -0.04 (0.2)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=11) | Placebo (N=10)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
left ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nausea (General disorders) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small exploratory study that may have been hindered due to lack of adequate power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No